CLINICAL TRIAL: NCT04399356
Title: Niclosamide for Patients With Mild to Moderate Disease From Novel Coronavirus (COVID-19)
Brief Title: Niclosamide for Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000605
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus; Treatment; Pill; Telehealth; Viral shedding
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Niclosamide

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: As all members of the Study Team will be blinded, Tufts Investigational Drug Services (IDS) will be unblinded and will dispense both the Niclosamide and placebo. The study intervention (Niclosamide) and placebo will be packaged and as indistinguishable as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Niclosamide (Active Comparator): Participants in the treatment arm will receive Niclosamide 2 grams orally on day 1 and daily for 6 more days (total 7 days of treatment)
  Interventions: Drug: Niclosamide; Other: Telehealth monitoring
- Control (Placebo Comparator): Participants in the control group will receive identical-appearing placebo by mouth in the same numbers of pills on day 1 and daily for 6 more days (total 7 days of treatment)
  Interventions: Drug: Placebo; Other: Telehealth monitoring

INTERVENTIONS:
Drug: Niclosamide — Participants in the treatment arm will receive Niclosamide 2 grams orally once daily for 7 days in addition to current standard of care treatment. Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 3, 7, 10, 14. Fecal samples will be collected for viral shedding as measured by PCR on days 3, 7, 10, 14, 21. A baseline fecal and oropharyngeal sample will be obtained on Day 1 prior to starting dosing of Niclosamide/ placebo.
  Arms: Niclosamide
Drug: Placebo — The collection of oropharyngeal samples will be observed by a Study Team member via the telehealth platform.
  Arms: Control
Other: Telehealth monitoring — In addition to Niclosamide or placebo treatments, all enrolled patients will be provided a home thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. The collection of oropharyngeal samples will be directly observed by a Study Team member via the telehealth platform.

SUMMARY:
This study will evaluate the antihelmintic drug, Niclosamide, as a potential treatment for mild to moderate coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
Niclosamide, which has potent antiviral activity against single-stranded RNA viruses including coronaviruses, was proposed as an antiviral during the Severe Acute Respiratory Syndrome (SARS) outbreak in 2002 and has activity including Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) where it was found to inhibit SARS coronavirus, SARS-CoV, in in vitro studies and similarly structured RNA viruses (both in vitro and in vivo). The investigators hypothesize that the antiviral activity of Niclosamide may be extended to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test by PCR
* No requirement of oxygen supplementation
* Ability to take oral medication

Exclusion Criteria:

* Known allergic reactions to any components of Niclosamide medication
* Participation in another trial or use of any experimental treatment for COVID-19, including chloroquine, hydroxychloroquine, remdesivir, and lopinavir/ritonavir
* Hospitalization or requirement of hospitalization at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry P Selker, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Cairns DM, Dulko D, Griffiths JK, Golan Y, Cohen T, Trinquart L, Price LL, Beaulac KR, Selker HP. Efficacy of Niclosamide vs Placebo in SARS-CoV-2 Respiratory Viral Clearance, Viral Shedding, and Duration of Symptoms Among Patients With Mild to Moderate COVID-19: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2144942. doi: 10.1001/jamanetworkopen.2021.44942. PMID 35138402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was among individuals reporting at Tufts Medical Center and Wellforce Network in Massachusetts for outpatient COVID-19 testing. The trial opened to accrual on October 1, 2020; the last participant enrolled on April 20, 2021.
Pre-assignment Details: Of 139 participants were assessed for eligibility, 73 met inclusion criteria and were randomized to treatment (66 participants were excluded: 23 did not meet inclusion criteria, 42 declined participation, 1 co-habited with a previously enrolled participant).
Groups:
- Niclosamide- Experimental Group: Participants received Niclosamide 2 grams by mouth daily for 7 days.
- Control Group: Participants received placebo using the same dosing schedule as Experimental Group
Period: Overall Study
Arm/Group | Niclosamide- Experimental Group | Control Group
Started | 36 | 37
Completed | 33 | 34
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Discontinued Niclosamide/ Placebo | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niclosamide | Control | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.82 (12.92) | 35.97 (13.27) | 36.39 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 24 | 32 | 56
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 26 | 27 | 53
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to Respiratory Viral Clearance
Description: Respiratory viral clearance is defined as the first day a participant's oropharyngeal (oral) sample result is negative, provided that none of the subsequent oral sample results are positive. We will calculate the time to clearance since Day 1.
Time Frame: Reduction in viral shedding as measured by oropharyngeal swab on days, 3, 7, 10, 14.
Population: We evaluated efficacy of niclosamide in shortening contagious period as determined by time to oropharyngeal viral clearance. Primary analysis was based on ITT population (all randomized participants). The cumulative probability of being in clearance in each randomization group was calculated using the Kaplan-Meier estimator. The cumulative probability of clearance at day 3 between the groups was calculated using a chi-square test based on a log(- log(·)) transformation for the survival function.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Niclosamide- Experimental Group | Control Group
Number analyzed (Participants) | 33 | 34
Days | 3.39 [1.88 to 4.91] | 3.44 [2.23 to 4.65]

2. Secondary Outcome: Time to Fecal Viral Clearance
Description: Reduction in fecal viral shedding as measured by fecal PCR on days, 3, 7, 10, 14 and 21. Fecal viral clearance is defined as the first day a participant's fecal sample result is negative, provided that none of the subsequent fecal sample results are positive; calculated as the time to clearance since Day 1.
Time Frame: Reduction in fecal viral shedding as measured by fecal PCR on days, 3, 7, 10, 14 and 21.
Population: We evaluated efficacy of niclosamide in shortening contagious period as determined by time to fecal viral clearance. Primary analysis was based on ITT population (all randomized participants). The cumulative probability of being in clearance in each randomization group was calculated using the Kaplan-Meier estimator. The cumulative probability of clearance at day 14 between the groups was calculated using a chi-square test based on a log(- log(·)) transformation for the survival function.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Niclosamide- Experimental Group | Control Group
Number analyzed (Participants) | 33 | 34
Days | 6.12 [3.51 to 8.73] | 5.77 [3.3 to 8.23]

3. Secondary Outcome: Number of Participants With Progression to Severe COVID-19 Disease
Description: Defined as 1) O2 saturation <92% on room air (in two consecutive measurements at least 2 hours apart) OR 2) requirement of hospitalization OR 3) need for artificial ventilation OR 4) death. 1) We will compare the proportion of participants who progressed to severe COVID disease between groups.
Time Frame: Day 1- 30
Population: Progression to Severe COVID
Measure: Count of Participants; unit: Participants
Arm/Group | Niclosamide- Experimental Group | Control Group
Number analyzed (Participants) | 33 | 34
Participants | 0 | 1

4. Secondary Outcome: Number of Days to Resolution of a Fever
Description: Mean time to fever resolution (symptom no longer reported).
Time Frame: Day 1-30
Population: The mean time to resolution of fever *symptom no longer reported)
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Niclosamide- Experimental Group | Control Group
Number analyzed (Participants) | 33 | 34
Days | 10.2 [1.86 to 18.54] | 3.6 [2.07 to 5.13]

ADVERSE EVENTS:
Time Frame: 30 days
Description: CTCAE V5.0
Arm/Group | Niclosamide- Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 5/33 | 12/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niclosamide- Experimental Group (N=33) | Control Group (N=34)
Skin rash (Skin and subcutaneous tissue disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 7

LIMITATIONS AND CAVEATS:
There was a precipitous and persistent decrease in the rate of COVID-19 diagnoses in spring and summer 2021 that decreased our enrollment pool. Additionally, as vaccination rates rose, our predetermined exclusion criteria of individuals vaccinated against SARS-CoV-2 limited those available for enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04399356/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT04399356/SAP_002.pdf